CLINICAL TRIAL: NCT02518087
Title: Increased Adsorption Membranes During Cardiopulmonary Bypass. a Randomized Controlled Trial to Evaluate Impact of OXiris® Membrane in Cardiac Surgery Associated Acute Kidney Injury
Brief Title: Increased Adsorption Membranes During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Germans TrÃ-es i Pujol de Badalona (Unknown); FundaciÃ³ Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Unknown); Baxter Healthcare Corporation (Industry); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, JOSE LUIS PEREZ FERNANDEZ, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIRAKI 02-2015
Record Dates: First submitted 2015-07-20; First posted 2015-08-07 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery Associated - Acute Kidney Injury; Systemic Inflammatory Response Syndrome; Acute Kidney Injury
Keywords: CPB; oXiris®; CSA-AKI; SIRS; Cytokines; LPS; AKI
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPB-oXiris® (Experimental): Non emergent cardiac surgery patients requiring expected CPB time > 90 minutes: double valve replacement or valve replacement plus coronary arterial bypass graft (CABG).
  Interventions: Device: oXiris®
- CPB-Standard (No Intervention): Non emergent cardiac surgery patients requiring expected CPB time > 90 minutes: double valve replacement or valve replacement plus coronary arterial bypass graft (CABG).

INTERVENTIONS:
Device: oXiris® — oXiris® membrane set is composed of a 1.5 m2 copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface and adhered heparin during set´s fabrication [oXiris® (Baxter Gambro)].
  Blood flow between 200-250 mL/min will be derivatised from the CPB circuit (arterial positive pressure line just after the oxygenator) into the PrismafleX eXeed™, so that it all flows thru the oXiris® membrane and returned to the CPB circuit into the venous reservoir just before the oxygenator. oXiris® membrane will be only employed for adsorption (neither convection nor diffusion will be performed) during all CPB time.
  Arms: CPB-oXiris®

SUMMARY:
Our project intends to reduce cardiac surgery associated - acute kidney injury (CSA-AKI) in non emergent patients with the use of an increased adsorption membrane (oXiris®) connected to the cardiopulmonary bypass (CPB) circuit, besides evaluating the inflammatory response by quantifying inflammatory mediators during and after cardiac surgery with CPB. Our study is a randomized and controlled multicentre trial that includes recruiting centres with a long experience in cardiac surgery with CPB.

The primary endpoint of the project is to evaluate the ability of oXiris® to reduce the incidence of CSA-AKI in patients undergoing non emergent cardiac surgery with an expected CPB time of more than 90 minutes (doble valve replacement or valve replacement plus coronary artery bypass graft). With the goal of reducing by 10% (from 25 to 15%) the risk of CSA-AKI during the first postoperative week a sample size of 340 patients has been calculated.

Secondary endpoints are two; first, to evaluate the effect of using oXiris® on survival, clinical course and removal capacity of cytokines and lipopolysaccharide (LPS) during and after CPB; and second, to assess the predictive value for CSA-AKI of some new biomarkers, such as uNAD (urinary nicotinamide adenine dinucleotide).

DETAILED DESCRIPTION:
The oXiris® set connection to CPB

* The PrismafleX eXeed™ II (Baxter) system control unit will be used to deliver CRRT and thus connected to the CPB circuit through the oXiris® set lines.
* Priming. For oXiris® set priming use 2 L of normal saline according to the software instructions.
* Connection. Using a three-way stopcock, oXiris® set must be connected to the arterial line just after the oxygenator to derive blood into the oXiris® set and then returned into the venous reservoir through the return line. No additional vascular access will be required to deliver treatments.
* Modality. The Slow Continuous Ultrafiltration modality (SCUF modality) must be selected with no pre-set ultrafiltration rate (ultrafiltration rate: 0 ml/hr). A blood flow between 200-300 mL/min was set in the PrismafleX eXeed™ II (blood was derived through the arterial positive pressure line just after the oxygenator) to be delivered into the oXiris® set and then returned into the venous reservoir through the return line.
* All treatments should be delivered after reaching full-flow CPB.
* CRRT flow, pressure and alarms will be controlled in the PrismafleX eXeed™ II screen, independently from CPB circuit.
* If CPB is stopped for any reason, then PrismafleX eXeed™ II should be stopped temporarily to avoid alarm warning and/or any harm to the patient.
* No additional anticoagulation method will be needed besides the systemic anticoagulation required for the cardiopulmonary bypass pumping.
* The return line clamp (blue clamp) should be adjusted to reach a slight positive return pressure in order to avoid low-pressure alarm warning.

PrismafleX eXeed™ II weaning instructions. 5-10 min before the end of CPB, start the blood-return procedure into the venous reservoir of the CPB using 1 L of normal saline. Connect the solution into the three-way stopcock. Subsequently, set PrismafleX eXeed™ II flow in 80-100 ml/min. Select STOP in the PrismafleX eXeed™ II screen. Adjust the three-way stopcock to allow saline to flow into the oXiris® set arterial line an restart PrismafleX eXeed™ II to return blood into the venous reservoir.

• Register all manoeuvres, changes and adjustments in software settings and any technical problem during the procedure.

oXiris® membrane will be only employed for adsorption (neither convection nor diffusion will be performed) during all CPB time. Using CPB flow, patient will not require venous catheter access neither changes in CPB normal settings.

oXiris® membrane set is composed of a 1.5 m2 copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface and adhered heparin during set´s fabrication [oXiris® (Baxter Gambro)].

All blood samples collected during study will be obtained from CPB circuit or central venous catheters (standard cardiac surgery protocol).

During all CPB time besides the ordinary cardiac surgery assistance team, a supplementary CRRT expert team will be present in those patients randomized to CPB-oXiris®.

Blood samples and all variables will be equally collected and registered in the control group (CPB-Standard) with no modifications from CPB standard practice.

Adverse events will be reported (in less than 24 hours if severe) to the sponsor centre to be properly evaluated. If the severe adverse event (SAE) is finally evaluated by the study board as related to the intervention arm, urgent notification to health authorities must proceed and study should be interrupted until further decision.

Investigators will warrant a correct protocol application. Study data will be reviewed by an external monitoring committee from the clinical assay research central unit (UCICEC - IDIBELL). Monitors will contrast registered data from the collection data form (CDF) with data from patients' medical record. All patients' medical records will be indefinitely saved in electronic format to be reviewed if necessary.

Efficacy Assessments:

1. Registered variables and follow-up. Renal function related parameters Plasma creatinine and urine output will be registered at baseline, prior to CPB, at ICU admission, 6 hours ,12 hours, 24h postCBP and every 24h during the first week after cardiac surgery in order to evaluate CSA-AKI based on KDIGO AKI criteria (KDIGO criteria Kidney inter., Suppl. 2012; 2: 1-138.) Urinary NAD (uNAD) will also be quantified at ICU admission. Renal function will be checked at hospital discharge.

   Inflammatory response parameters Interleukin-1β (IL-1β), tumor necrosis factor alpha (TNF-α), monocyte chemotactic protein-1 (MCP-1), interleukin-4 (IL-4), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-18 (IL-18), complement 5a (C5a), high mobility binding protein 1 (HMBP-1), RANTES, GRO-alpha, leukocytes count, lactate, D-dimer, free plasma hemoglobin, HO-1, free iron and Lipopolysaccharide (LPS) levels will be determined in plasma.These determinations will be measured baseline (0 hours), and at times T1 (at the end of CPB), T2 (ICU admission) and T3 (24 hours after ICU admission).

   Ordinary laboratory parameters Plasmatic urea, potassium, albumin, magnesium, phosphate, glucose, sodium, chloride, AST, ALT, blood cell count and coagulation times will be determined following the ordinary cardiac surgery protocol (every 8 hours during the first 24h).

   Clinical and respiratory parameters Hemodynamic and respiratory parameters will be registered every hour. Arterial and venous blood gases with arterial lactate will be determined every 8 hours during the first 24 hours. Temperature, heart rate, arterial blood pressure (systolic, diastolic, and mean), central venous pressure, vasopressor and/or inotrope dose will be registered during surgery and at ICU according to standard protocol.

   Demographic and clinical record data Age, gender, weight, height, relevant clinical records, previous or chronic medication, type of cardiac surgery, surgery times, time on CPB, surgical complications, blood transfusions during and after surgery, prognostic scores (SOFA, APACHE II and SAPS II), ICU stay, hospital stay. Clinical outcome (survival at discharge, 28 and 90 days) and renal outcome (renal function, and RRT requirements).
2. Techniques. Lipopolysaccharide (LPS) LPS plasmatic concentration will be measured using an Limulus amebocyte lysate (LAL) test (Levin, J, et al. Thrombosis Et Diathesis Haemorrhagica. 1968; 19:186). This technique is performed when LAL proteolytic factors are activated by LPS. Life Technologies kit will be used for this (Thermo Fischer Scientific).

NAD Urinary and blood levels of NAD will be determined at 0 hours and at times T1 (end of CPB), T2 (ICU admission), and T3 (24 hours after ICU admission) applying multiplexed mass spectrometry techniques.

Cytokine analysis IL-1, IL-4, IL-6, IL-8, IL-10, IL-18, TNFα, MCP-1, HMBP-1, RANTES, GROα quantification will be performed with multiplex new technology. MILLIPLEX (Millipore) magnetic balls system will be used.

LPS, NAD, and Cytokine analysis will be all performed after completing recruitment and in the meantime all samples will be safely stored at -70°C.

Statistical Methods (for analyzing primary & secondary endpoints):

Statistical analysis will be done by the statistics investigator who won't have any role in patient selection, randomization, or follow up. SPSS v. 20.0 for statistical analysis will be used. Variable distribution will be studied and logarithmic transformation will be used on those variables that don't present normal distribution, presumably cytokine and LPS levels. Univariate analysis comparing clinical, demographic, biochemical, metabolic, hemodynamic and respiratory baseline variables between both arms (CPB-oXiris® and CPB-Standard), will be done with two-tailed t test for continuous variables and chi-square test for categorical variables.

Variables determined several times (T0, T1, T2, T3) will be analysed using a one-way repeated measures ANOVA test in order to demonstrate differences between both arms. Multivariate analysis will be completed to control those clinically relevant confounding variables as well as to discover baseline differences. According to hypothesis and to the dependent variable on study investigators will use a survival analysis (to study CSA-AKI within the first week postsurgery) with a Cox regression model, or a hierarchic multiple linear regression model when the dependent variable is continuous (for example, uNAD). Arm intervention (CPB-oXiris®, CPB-Standard) will be considered as the main independent variable adding other control independent variables.

As the study is measuring cytokine and LPS levels in four different moments (T0, T1, T2, T3), in order to maximize statistical power and reduce control variables number, the area under the curve (AUC) will be calculated for every cytokine and LPS during the first 24 hours. Due to this statistical maneuver investigators will obtain a continuous variable that represents each cytokine-LPS level during the biochemical study period (24 hours). To evaluate if the arm intervention improvement in terms of efficacy and safety could be related to cytokine and/or LPS levels during the first 24 hours, a mediation complementary analysis will be performed considering cytokine-LPS (represented by AUC) as a mediator between the independent variable (intervention arm) and the effect we study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 18 years old.
* Non emergent cardiac surgery patients requiring expected CPB time > 90 minutes: double valve replacement or valve replacement plus coronary arterial bypass graft (CABG).
* Written informed consent from patient or legal surrogates.

Exclusion Criteria:

* Immunosuppressive treatment or steroids (prednisone > 0.5 mg/kg/day or equivalent).
* Autoimmune disorder.
* Transplant receptor.
* Advanced Chronic Kidney Disease (CKD 4 or 5).
* Renal replacement therapy in the last 90 days.
* Documented intolerance to study device.
* Inclusion in other ongoing study within the last 30 days.
* Pregnancy.
* Coexisting illness with a high probability of death (inferior to 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Non presence of CSA-AKI within the first 7 days after cardiac surgery. | 7 days
  Participants who underwent cardiac surgery with no CSA-AKI within the first 7 days after cardiac surgery. CSA-AKI will be defined as at least AKI stage≥1 (according to AKI KDIGO classification) during the first 7 days of cardiac surgery. Patients with previous mild chronic kidney disease (CKD) will also be classified as CSA-AKI according to changes of creatinine respect to baseline creatinine or urine output decrease within the first 7 days after cardiac surgery.

SECONDARY OUTCOMES:
90 day survival after cardiac surgery. | 90 days
  90 day survival evaluation after cardiac surgery.
ICU length of stay after cardiac surgery. | Participants will be followed for the duration of ICU stay, an expected average of 2 days.
  ICU length of stay evaluation after cardiac surgery.
Cytokine circulatory levels during CPB and up to 24 hours after surgery. | First 24 hours after cardiac surgery.
  Cytokine circulatory levels during CPB and up to 24 hours after surgery. Cytokine removal: IL-1, IL-6, IL-8, IL-10, IL-18, TNFα, MCP-1, HMBP-1, RANTES, and GROα levels will be determined in plasma.
  Determinations will be measured baseline (0hours), and at T1 (CPB end), T2 (ICU admission), and T3 (24hours).
Urinary and blood levels of NAD values after cardiac surgery. | First 24 hours after cardiac surgery.
  Urinary and blood levels of NAD will be at measured baseline (0hours), and at T1 (CPB end), T2 (ICU admission), and T3 (24hours).
Composite Creatinine and Urine output after cardiac surgery. | 7 days after cardiac surgery.
  Renal function in terms of creatinine and urine output will be registered every 24h after cardiac surgery up to the first week. KDIGO AKI score will be calculated according to these two items.
Hospital length of stay after cardiac surgery. | Participants will be followed for the duration of hospital stay, an expected average of 1 week.
  Hospital length of stay evaluation after cardiac surgery.
LPS circulatory levels during CPB and up to 24 hours after surgery. | First 24 hours after cardiac surgery.
  Lipopolysaccharide (LPS) removal: LPS levels will be determined in plasma. Determinations will be measured baseline (0hours), and at T1 (CPB end), T2 (ICU admission), and T3 (24hours).

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabater Riera, MD PhD, Principal Investigator — Hospital Universitari de Bellvitge; Xosé L Perez-Fernandez, MD, Principal Investigator — Hospital Universitari de Bellvitge; Kathleen D Liu, MD PhD, Study Chair — University California San Francisco
Locations (3):
- Spain (3):
  - Hospital German Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Statement Data Additional Information: NCT02518087 Data available: Yes Data types: Deidentified participant data How to access data: xose74@gmail.com When available: With publication Supporting Documents Document types: Statistical/analytic code, Informed consent form How to access documents: xose74@gmail.com When available: With publication Additional Information Who can access the data: researchers whose proposed use of the data has been approved Types of analyses: Specified purpose Mechanisms of data availability: Signed data access agreement
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Perez-Fernandez X, Ulsamer A, Camara-Rosell M, Sbraga F, Boza-Hernandez E, Moret-Ruiz E, Plata-Menchaca E, Santiago-Bautista D, Boronat-Garcia P, Gumucio-Sanguino V, Penafiel-Munoz J, Camacho-Perez M, Betbese-Roig A, Forni L, Campos-Gomez A, Sabater-Riera J; SIRAKI02 Study Group. Extracorporeal Blood Purification and Acute Kidney Injury in Cardiac Surgery: The SIRAKI02 Randomized Clinical Trial. JAMA. 2024 Nov 5;332(17):1446-1454. doi: 10.1001/jama.2024.20630. PMID 39382234